CLINICAL TRIAL: NCT04078971
Title: Effects of a Very Low Carbohydrate Ketogenic Diet on Body Composition, Muscle Strength, Muscle Area, Metabolism and Performance in Semi-professional Soccer Players
Brief Title: Effects of Ketogenic Diet on Body Composition and Performance in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Paoli (Other)
Responsible Party: Sponsor-Investigator, Antonio Paoli, Professor, University of Padova
Organization: University of Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KDsoccer
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Athletic Performance
Keywords: ketogenic diet; western diet; soccer; sport performance; muscle mass; body composition
MeSH Terms: interventions — Diet, Western; Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: It is single blind, parallel arms study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Treatment and control were masked with A and B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Experimental): Ketogenic diet: less than 30 g/day of carbohydrate. Subjects can eat beef, veal, poultry, fish, raw and cooked vegetables without restriction, cold cuts such as dried beef, eggs and seasoned cheese (parmesan), ketogenic pasta (selected with a ketogenic ratio of 4:1), fruits with the lowest glycemic index (blueberry, raspberry), raw nuts and seeds, ghee butter, plant oils and fats from avocado, coconut and olives
  Interventions: Other: ketogenic diet
- Western diet (Active Comparator): The western diet (WD) is composed mainly of whole cereals (spelt, rye, oat) and pseudo-cereals (buckwheat, quinoa, amaranth), whole grain pasta, potatoes, meet, fish, vegetables, fruit, legumes, olive oil, milk and red wine (at most 1 glass per day). It ensure a constant energy and macronutrient balance: protein 1.8g x Kg-1 x body weight-1 x day-1, (30%), fats 20-25% and carbohydrate 50-55%.
  Interventions: Other: Western diet

INTERVENTIONS:
Other: Western diet — Subjects in this intervention will follow a normal western diet
  Arms: Western diet
Other: ketogenic diet — Subjects in this group will follow a low carbohydrate ketogenic diet
  Arms: Ketogenic diet

SUMMARY:
A ketogenic diet (KD) is a nutritional approach, usually adopted for weight loss, that restricts daily carbohydrates under 30 g/day. KD showed contradictory results on sport performance, whilst no data are available on team sports. The investigators will investigate the influence of a KD on different parameters in soccer players

DETAILED DESCRIPTION:
Sixteen semi-professional soccer players will be randomly assigned to a ketogenic diet (KD n=8) or to a western diet (WD n=8). Diets contain the same amount of protein (1.8g/Kg body weight/day). Body weight and body composition will be measured by dual energy x-ray absorptiometry (DXA) and bioelectrical impedance analysis (BIA). Resting energy expenditure (REE), respiratory exchange ratio (RER), cross sectional area (CSA) and isometric muscle strength of quadriceps, counter movement jump (CMJ) and yoyo intermittent recovery test will be measured.

ELIGIBILITY:
Inclusion Criteria

* semiprofessional soccer players
* male

Exclusion Criteria:

* body fat percentage over 32%, (determined via dual energy X-ray absorptiometry DEXA),
* cardiovascular,
* respiratory, gastrointestinal,
* thyroid or any other metabolic diseases,
* weight change more than 2 Kg over the last month,
* adherence to special diets,
* use of nutritional supplements (except a daily multivitamin-mineral)
* use of medication to control blood lipids or glucose and goal-keepers.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Fat body mass | 4 weeks
  Body composition with DEXA: we measure body fat mass in grams.
lean body mass | 4 weeks
  Body composition with DEXA: we measure lean body mass in grams.
Visceral Adipose tissue (VAT) | 4 weeks
  Body composition with DEXA: VAT in grams
Total body water | 4 weeks
  We will use a BIA to calculate totally body water and intracellular and extracellular water in liters

SECONDARY OUTCOMES:
resting energy expenditure (REE) | 4 weeks
  Measured through gas analyzer in ml/02/kg min
respiratory ratio (RR) | 4 weeks
  Measured through gas analyses (ratio between CO2 and O2)
specific performance | 4 weeks
  Yoyo intermittent recovery test level 1: in seconds
lower limb power | 4 weeks
  squat jump test: height of the jump in cm
quadriceps muscle area | 4 weeks
  muscle area measured in cm2 through ultrasound
quadriceps muscle thickness | 4 weeks
  muscle thickness measured cm through ultrasound
quadriceps strength | 4 weeks
  isometric contraction measured in N, the normalized per muscle area (N x cm2)
quadriceps strength per area | 4 weeks
  the strength of isometric contraction (outcome 10) normalized per muscle area (Outcome 7). Expressed as (N x cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
Raw data of outcomes on request

REFERENCES:
- [Background] Rubini A, Bosco G, Lodi A, Cenci L, Parmagnani A, Grimaldi K, Zhongjin Y, Paoli A. Erratum to: Effects of Twenty Days of the Ketogenic Diet on Metabolic and Respiratory Parameters in Healthy Subjects. Lung. 2017 Feb;195(1):155. doi: 10.1007/s00408-016-9958-0. No abstract available. PMID 27803969
- [Background] Paoli A, Bianco A, Grimaldi KA. The Ketogenic Diet and Sport: A Possible Marriage? Exerc Sport Sci Rev. 2015 Jul;43(3):153-62. doi: 10.1249/JES.0000000000000050. PMID 25906427
- [Background] Paoli A, Grimaldi K, D'Agostino D, Cenci L, Moro T, Bianco A, Palma A. Ketogenic diet does not affect strength performance in elite artistic gymnasts. J Int Soc Sports Nutr. 2012 Jul 26;9(1):34. doi: 10.1186/1550-2783-9-34. PMID 22835211
- [Derived] Antonio Paoli A, Mancin L, Caprio M, Monti E, Narici MV, Cenci L, Piccini F, Pincella M, Grigoletto D, Marcolin G. Effects of 30 days of ketogenic diet on body composition, muscle strength, muscle area, metabolism, and performance in semi-professional soccer players. J Int Soc Sports Nutr. 2021 Sep 16;18(1):62. doi: 10.1186/s12970-021-00459-9. PMID 34530857